CLINICAL TRIAL: NCT01776957
Title: Preventing Repeat Abortion: Is the Immediate Insertion of Intrauterine Devices Post-abortion a Cost-effective Option Associated With Fewer Repeat Abortions? Findings From 2005-2006 Data
Brief Title: Post Abortion IUD & Recurrent Abortion 2005-2006
Status: Terminated | Type: Observational
Why Stopped: This study is a retrospective chart review study, not a clinical trial.
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Wendy Norman, Principle Investigator, University of British Columbia
Other Study IDs: H12-00829
Record Dates: First submitted 2013-01-21; First posted 2013-01-28 (Estimated); Last update posted 2018-05-04 (Actual); Status verified 2018-05

CONDITIONS: Induced Abortion
Keywords: Abortion rate; Intrauterine device
MeSH Terms: interventions — Intrauterine Devices

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- IUD: Repeat abortion rate in women receiving IUDs immediately post-abortion
  Interventions: Device: Device: Intrauterine device (IUD)

INTERVENTIONS:
Device: Device: Intrauterine device (IUD) — Women choosing to have an intrauterine device (IUD) inserted immediately post-abortion

SUMMARY:
The rate of repeat abortions will be lowest in those women who choose immediate insertion of an IUD post-abortion versus those who immediately choose oral contraceptive pills and those who indicate all other contraceptive choices including no contraception The provision by the health system of IUDs for immediate insertion will result in the lowest health system costs.

DETAILED DESCRIPTION:
The investigators intend to demonstrate whether there are statistically significant differences in the rates of repeat abortions between three groups: 1. women choosing to have an intrauterine device (IUD) inserted immediately post-abortion, 2. those choosing to begin oral contraceptives immediately post-abortion, and 3. all other choices for post abortion contraception including those stating an intention to obtain contraceptives at a later time or from an alternate location or to use no contraception. This data will then be used to conduct a cost-effectiveness analysis of health system provision for cost-free IUDs post-abortion. Thus, if providing a free IUD immediately post-abortion significantly reduces the rate of repeat abortions, it may be more cost- effective for health system services to provide free IUDs at abortion clinics than to field the costs associated with a higher rate of repeat abortions.

The researchers will conduct a retrospective observational cohort study by chart review. The researchers propose to review the charts of women undergoing abortions between January 1, 2005 and December 31, 2006 at Kelowna General Hospital's Women's Services Clinic. The researchers will record the following data from each chart: age, parity, gestational age, date of index therapeutic abortion (TA), dates of subsequent TAs, contraception used at the time of the index conception, contraceptive method chosen post-abortion, and outcome of follow-up at two weeks, such as expulsion of IUD. The researchers will also record the recurrent pregnancy rates.

ELIGIBILITY:
Inclusion Criteria:

* Female resident of Interior Health region seeking an abortion between January 1, 2005 and December 31, 2006

Exclusion Criteria:

* Women undergoing abortions for fetal genetic abnormalities

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female resident of Interior Health region seeking an abortion
Sampling Method: Non-Probability Sample
Enrollment: 1308 (Actual)
Dates: Start 2012-07; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
The proportion of repeat abortions at five years from the index abortions | 5 years

SECONDARY OUTCOMES:
Correlation of repeat and index abortions with obstetrical, demographic and contraceptive history factors. | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Norman, Dr., Principal Investigator — University of British Columbia